CLINICAL TRIAL: NCT02434744
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of KD026 in Combination With Metformin in Subjects With Type 2 Diabetes Mellitus
Brief Title: Study of KD026 in Combination With Metformin in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Response Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KD026-201
Record Dates: First submitted 2015-04-28; First posted 2015-05-05 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 6-(4'-trifluoromethyl-6-methoxybiphenyl-2-ylcarboxamido)-1,2,3,4-tetrahydroisoquinoline-2-carboxylic acid phenyl ester; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 100 mg KD026 BID (Experimental): 100 mg KD026 twice a day (BID) in combination with Metformin for 12 weeks
  Interventions: Drug: KD026; Drug: Metformin
- Cohort 2 150 mg KD026 BID (Experimental): 150 mg KD026 BID in combination with Metformin for 12 weeks
  Interventions: Drug: KD026; Drug: Metformin
- Cohort 3 200 mg KD026 BID (Experimental): 200 mg KD026 BID in combination with Metformin for 12 weeks
  Interventions: Drug: KD026; Drug: Metformin
- Cohort 4 100 mg KD026 TID (Experimental): 100 mg KD026 three times a day (TID) in combination with Metformin for 12 weeks
  Interventions: Drug: KD026; Drug: Metformin
- Cohort 1 Placebo (Placebo Comparator): Matched Placebo Dose BID in combination with Metformin for 12 weeks
  Interventions: Drug: Placebo; Drug: Metformin
- Cohort 2 Placebo (Placebo Comparator): Matched Placebo Dose BID in combination with Metformin for 12 weeks
  Interventions: Drug: Placebo; Drug: Metformin
- Cohort 3 Placebo (Placebo Comparator): Matched Placebo Dose BID in combination with Metformin for 12 weeks
  Interventions: Drug: Placebo; Drug: Metformin
- Cohort 4 Placebo (Placebo Comparator): Matched Placebo Dose TID in combination with Metformin for 12 weeks
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: KD026 — Dosed in combination
  Other Names: SLx-4090
  Arms: Cohort 1 100 mg KD026 BID; Cohort 2 150 mg KD026 BID; Cohort 3 200 mg KD026 BID; Cohort 4 100 mg KD026 TID
Drug: Placebo — Dosed in combination
  Arms: Cohort 1 Placebo; Cohort 2 Placebo; Cohort 3 Placebo; Cohort 4 Placebo
Drug: Metformin — Drug prescribed by each subject's prescribing physician

SUMMARY:
This study will compare the safety, tolerability and efficacy of the combination of KD026 and metformin compared to placebo and metformin on improving glycemic control in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes, with finger stick HbA1c ≥ 7.0% and ≤ 11.0% at screening visit, and HbA1c via venipuncture ≥ 7.0% and ≤ 11.0 % at the Qualification visit
* Have been on metformin for at least 12 weeks prior to screening visit and the metformin dose is not expected to change during the 4-week run-in period
* Have a BMI of ≥ 27 kg/m2 and ≤ 45 kg/m2
* Men, post-menopausal women (defined as not having a menstrual period for at least 1 year), surgically sterile women (for at least 1 year), or women of childbearing potential with a negative pregnancy test within the last 24 hours
* Women of childbearing potential and men whose partners are of childbearing potential must agree to use two forms of accepted methods of contraception during the course of the study and for 1 month after their last dose of study drug. Effective birth control includes (a) IUD plus one barrier method; (b) on stable doses of hormonal contraception for at least 3 months (eg, oral, injectable, implant, transdermal) plus one barrier method; (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or (d) a vasectomized partner

Exclusion Criteria:

* Have type 1 diabetes
* Taking antidiabetic medications other than or in addition to metformin
* Have fasting plasma glucose > 270 mg/dL at screening visit
* Have a serum creatinine ≥1.7 mg/dL or glomerular filtration rate <60 mL/min at screening visit
* Have a history of diabetic retinopathy
* Uncontrolled high blood pressure
* Have a history of chronic liver disease and/or alanine transaminase (ALT) or aspartate transaminase (AST) >2.0 × the upper limit of normal (ULN) at screening visit.
* Have a history of a malignant cancer (other than basal cell, localized cervical, or squamous cell carcinoma of the skin that has been removed)
* Have a history or presence of gastrointestinal (GI) disease or major gastrointestinal surgery that, in the opinion of the investigator, could interfere with drug absorption
* Currently using any of prohibited medications that cannot be stopped
* Abuse alcohol (defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units [1 unit is equivalent to a half pint of beer, 1 serving of hard liquor, or one glass of wine]
* History or presence of drug abuse according to Diagnostic and Statistical Manual of Mental Disorders V (DSM-V) criteria within the 2 years prior to screening visit
* Have a 12-lead ECG at screening visit that, in the opinion of the investigator, have abnormalities that may compromise safety in this study, including a QTc(F) interval (QT interval data corrected using Fridericia's formula) of > 450 msec
* Have a clinically significant abnormal laboratory result including thyroid-stimulating hormone (TSH) >1.5 × ULN at screening visit
* Have a positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody/virus (HCV) or human immunodeficiency virus (HIV) antibodies at screening visit or a documented history of a positive result
* Pregnant or lactating woman
* Previously received KD026 (formerly named SLx-4090)
* Participated in a trial with any investigational drug within 4 weeks prior to screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of Subjects Experiencing Adverse Events as a Measure of Safety, Tolerability, and Efficacy | 12 Weeks
  To assess the safety, tolerability, and efficacy (as measured by a 0.5%-1.5% decrease of HbA1c) of different dosages and dosing regimens of a combination of KD026 and metformin compared to placebo and metformin when administered for 3 months to subjects with type 2 diabetes mellitus

SECONDARY OUTCOMES:
Changes in Fasting Plasma Glucose (FPG) | 12 Weeks
  To assess changes in fasting plasma glucose from baseline to Week 12
Changes in Insulin | 12 Weeks
  To assess changes in insulin from baseline to Week 12
Changes in HOMA-IR | 12 Weeks
  To assess changes in Homeostasis Model Assessment - Insulin Resistance (HOMA-IR) from baseline to Week 12
Changes in Body Weight | 12 Weeks
  To assess changes in body weight
Changes in AUC | 12 Weeks
  To assess the 6-hour time curve (AUC) for post prandial triglycerides and glucose.
Changes in Lipids | 12 Weeks
  To assess changes in total cholesterol, LDL-C, HDL-C, non-HDL-C, VLDL-C, and triglyceride levels
Changes in Blood Pressure | 12 Weeks
  To assess changes, if any, in baseline blood pressure associated with metabolic syndrome
Changes in Waist Circumference | 12 Weeks
  To assess changes, if any, in baseline waist circumference associated with metabolic syndrome
Changes in Body Mass Index (BMI) | 12 Weeks
  To assess changes, if any, in baseline measures of BMI associated with metabolic syndrome
Changes in Plasma Levels of KD026 | 12 Weeks
  To assess plasma levels of KD026 in all subjects
Changes in Serum Levels of Non-Esterified Free Fatty Acids | 12 Weeks
  To assess the change in serum levels of non-esterified free fatty acids from baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Axis Clinical Trials, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Infosphere Clinical Research, Inc, West Hills, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Med Research of Florida, LLC, Miami, Florida
  - High Point Clinical Trials Center, High Point, North Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Trial Network, Houston, Texas
  - Clinical Research Associates of Tidewater, Norfolk, Virginia